CLINICAL TRIAL: NCT01014637
Title: A Multicentre, Randomized, Controlled Study of the Efficacy, Safety and Cost-effectiveness of a Sequential Therapy With RV4104A Ointment, Ciclopiroxolamine Cream and Ciclopirox Film-forming Solution Compared With Amorolfine Nail Lacquer Alone for the Treatment of Dermatophytic Onychomycosis (Toenail) Without Matrix Involvement
Brief Title: Efficacy, Safety and Cost-effectiveness of a Sequential Therapy With RV4104A Ointment, Ciclopiroxolamine Cream and Ciclopirox Film-forming Solution Compared With Amorolfine Nail Lacquer in Dermatophytic Onychomycosis
Acronym: ONICO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Collaborators: Quanta Medical (Industry)
Responsible Party: Anne-Marie Schmitt, MD, Pierre Fabre Dermo Cosmetiques
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV4104A 2008 548
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Onychomycosis
Keywords: Dermatomycoses; Infection; Mycoses; Nail diseases; Ski diseases; Skin diseases/infectious
MeSH Terms: conditions — Onychomycosis; Dermatomycoses; Infections; Mycoses; Nail Diseases; Cellulitis | interventions — amorolfine; Antifungal Agents; Ciclopirox; Keratolytic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amorolfine 5% (Active Comparator)
  Interventions: Drug: Amorolfine (Antifungal)
- RV4104A-cylcopiroxolamine-ciclopirox (Experimental)
  Interventions: Drug: RV4104A, Ciclopiroxolamine, Cyclopirox (Keratolytic Agents/Antifungal)

INTERVENTIONS:
Drug: Amorolfine (Antifungal) — Treatment with Amorolfine for 36 weeks
  Other Names: Loceryl
  Arms: Amorolfine 5%
Drug: RV4104A, Ciclopiroxolamine, Cyclopirox (Keratolytic Agents/Antifungal) — Initial treatment with RV4104A ointment for 3 weeks, followed by treatment with ciclopiroxolamine 1% cream for 8 weeks and by cyclopirox 8% film-forming solution for 25 weeks.
  Other Names: RV4104A ointment; Mycoster 1%; Mycoster 8%
  Arms: RV4104A-cylcopiroxolamine-ciclopirox

SUMMARY:
The purpose of the study is to evaluate and compare the efficacy of the sequential association RV4104A ointment followed by ciclopiroxolamine 1% cream and ciclopirox 8% film-forming solution versus amorolfine 5% nail lacquer alone in the treatment of patients with dermatophytic onychomycosis (toenail) without matrix involvement.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of distal-lateral or lateral subungual onychomycosis of one great toenail (the target nail) without matrix involvement
* Target nail plate showing between 25% and 60% of clinically infected area
* Patient must have at least 2 mm of unaffected proximal target nail area
* Target nail infection due exclusively to a dermatophyte (from positive fungal culture as reported by the central mycological laboratory)
* Female patient of childbearing potential must use an efficient contraceptive method for at least 2 months prior to screening visit
* Female patient of childbearing potential must have a negative urinary pregnancy test at the screening visit

Exclusion Criteria:

* Patient with more than 3 affected nails
* Patient with onychomycosis with matrix involvement
* Patient with psoriasis, lichen planus or other abnormalities that could result in clinically abnormal toenail(s)
* Patient with moccasin-type tinea pedis
* Patient who has received systemic antifungal therapy or any topical antifungal therapy applied to the toenails within 3 months prior to screening visit
* Patient with known hypersensitivity to investigational products' ingredient(s)
* Patient who is currently participating or who has participated in another clinical study within 4 weeks prior to screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate and compare the efficacy of the sequential association RV4104A ointment-ciclopiroxolamine 1% cream-ciclopirox 8% film-forming solution versus amorolfine 5% nail lacquer alone in dermatophytic onychomycosis (toenail) without matrix involvement | Day 336

SECONDARY OUTCOMES:
To evaluate and compare the local tolerability of the sequential association RV4104A-ciclopiroxolamine-ciclopirox versus amorolfine 5% alone in the treatment dermatophytic onychomycosis (toenail) without matrix involvement | Day 21, Day 77, Day 156, Day 262
To evaluate and compare the cost-effectiveness of the sequential association RV4104A ointment-ciclopiroxolamine 1% cream-ciclopirox 8% film-forming solution vs amorolfine 5% alone in the treatment of dermatophytic onychomycosis without matrix involvement | Day 336
To evaluate and compare the clinical cure of the sequential association RV4104A ointment-ciclopiroxolamine-ciclopirox 8 versus amorolfine alone in the treatment dermatophytic onychomycosis (toenail) without matrix involvement | Day 77, Day 168, Day 252
Averse Events Reporting | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Carle PAUL, Professor, Principal Investigator — Hopital Purpan
Locations (7):
- France (7):
  - Cabinet Médical, Argenteuil
  - Cabinet Médical, Brest
  - Cabinet Medical, Cholet
  - Cabinet Médical, Martigues
  - Cabinet Médical, Nice
  - Cabinet Médical, Toulouse
  - Hopital Purpan, Toulouse